CLINICAL TRIAL: NCT06755034
Title: Stabilizing Mandibular Overdentures With a Single Implant Placed in the Canine Region of the Preferred Chewing Side Compared to the Midline Single-implant Overdenture Treatment Concept: an RCT With 5 Years of Follow-up
Brief Title: Stabilizing Mandibular Overdentures With a Single Implant Placed in the Canine Region of the Preferred Chewing Side
Acronym: c-SIMO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Frauke Müller (Other)
Responsible Party: Sponsor-Investigator, Frauke Müller, Professor, Head of Division, University of Geneva, Switzerland
Organization: University of Geneva, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DGPA_2024_02
Record Dates: First submitted 2024-12-15; First posted 2025-01-01 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Completely Edentulous Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- c-SIMO (Experimental): Placement of an implant in the mandibular canine area and using it to stabilize a pre-existing mandibular complete denture.
  Interventions: Device: c-SIMO
- m-SIMO (Active Comparator): Placement of an implant in the midline of the mandible and using it to stabilize a pre-existing mandibular complete denture.
  Interventions: Device: m-SIMO

INTERVENTIONS:
Device: c-SIMO — Placement of an implant in the mandibular canine area and using it to stabilize a pre-existing mandibular complete denture.
  Arms: c-SIMO
Device: m-SIMO — Placement of an implant in the midline of the mandible and using it to stabilize a pre-existing mandibular complete denture.
  Arms: m-SIMO

SUMMARY:
The investigators are evaluating the use of a single implant to stabilize complete dentures in the lower jaw, in the canine region of the preferred chewing side. They are conducting this study to determine whether this treatment concept gives satisfactory results, and how it compares with the standard position in the center of the lower jaw.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed by the subject
* Age ≥ 60 years
* Edentulous and wearing sufficient complete maxillary and mandibular dentures or ones that can be rendered sufficient via a reline and/or renewal of the prosthetic teeth
* Healed edentulous mandible (minimum 6-8 weeks since last extraction in the anterior zone (4-4) and one year in the posterior zone (5-8))
* Physical status ASA1 and ASA2

Exclusion Criteria:

* Contraindications to the medical devices used, e.g. known hypersensitivity or allergy
* Vulnerable subjects
* Enrollment of the investigator, his/her family members, employees and other dependent persons
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to perform adequate oral hygiene
* Inability to follow the procedures of the investigation, e.g. due to language problems, psychological disorders, dementia, Parkinson etc. of the subject (Dementia: clock-drawing test score ≤ 5)
* Surgical risk factors such as, but not limited to, uncontrolled diabetes, immunosuppression, radiation, chemotherapy, or antiresorptive medication (ex. Bisphosphonates)
* Heavy smoking habit: >20 cig/d
* Reported severe bruxism or clenching habits, clinically present oro-facial pain
* Depression: Geriatric Depression Scale > 9
* Xerostomia: SSFR ≤ 0.7ml/min
* Ridge dimensions <6 mm (width) by 10 mm (height) in the canine or midline area
* Ridge defects requiring bone augmentation procedures

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2031-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
OHIP-EDENT | From baseline to 5-year follow-up
  Oral health-related quality of life questionnaire
DSI | From baseline to 5-year follow-up
  Denture Satisfaction Index (questionnaire)

SECONDARY OUTCOMES:
Preferred chewing side | From baseline to 5-year follow-up
  Asymmetry Index
Chewing efficiency | From baseline to 5-year follow-up
  two-color mixing ability test
Occlusal analysis | From baseline to 5-year follow-up
  Dental Prescale System
Plaque index | From implant loading to 5-year follow-up
  modified Plaque Index (modPI)
Bleeding on probing | From implant loading to 5-year follow-up
  modified Bleeding Index (modBI)
Pocket probing depth | From implant loading to 5-year follow-up
  Peri-implant probing depth
Keratinized peri-implant tissues | From implant loading to 5-year follow-up
  Measurement of the keratinized tissue around implants
Prosthodontic assessment | From implant loading to 5-year follow-up
  Number of prosthetic complications
Peri-implant bone height | From implant loading to 5-year follow-up
  Measured on radiographs

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Maniewicz, Principal Investigator — University of Geneva; Frauke Müller, Study Director — University of Geneva
Locations (1):
- University Clinics of Dental Medicine, University of Geneva, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No